CLINICAL TRIAL: NCT01217840
Title: The Effect of Vitamin D on Cytokines and Cardiometabolic Risk in Obese Adolescents
Brief Title: Effect of Vitamin D Supplementation on Inflammation and Cardiometabolic Risk Factors in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Laura K Bachrach, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-10012010-6989; 18885 (Other: Stanford IRB)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Adolescents, Vitamin D
MeSH Terms: conditions — Obesity | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D (Experimental): Subjects were assigned to receive two observed doses of vitamin D2 (150,000 IU ergocalciferol, Barr Laboratories and Winthrop (Sanofi-Aventis)), given at baseline and 12 weeks. Capsules were packaged by the hospital's clinical trial pharmacist and were administered by study staff blinded to group assignments.
  Intervention: Height, weight, and BMI were obtained at baseline, 12 weeks and 24 weeks
  Interventions: Drug: Drisdol (Ergocalciferol) Vitamin D2
- Placebo (Placebo Comparator): Subjects were assigned to receive two observed doses of placebo, given at baseline and 12 weeks. Capsules were packaged by the hospital's clinical trial pharmacist and were administered by study staff blinded to group assignments. Height, weight, and BMI were obtained at baseline, 12 weeks and 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drisdol (Ergocalciferol) Vitamin D2 — Ergocalciferol 150,000 IU every 12 weeks for total of 24 weeks.
  Arms: vitamin D
Drug: Placebo — Placebo pill - 3 pills every 12 weeks for total of 24 weeks
  Arms: Placebo

SUMMARY:
Large studies of children show that over half of the children in the United States of America do not have enough vitamin D stored in their bodies. In children who are overweight or obese, the percentage of children who do not have enough vitamin D is even higher.

Vitamin D is essential for the body to maintain normal calcium levels and strong bones. Recent research shows that through the actions of inflammatory markers, levels in the blood that measure inflammation in the body, vitamin D plays many other important roles in the body like helping to regulate the immune system, blood sugar levels, blood pressure, and body fat.

The purpose of this study is to determine the effect of vitamin D supplementation on inflammatory markers in obese and overweight adolescents. As a secondary goal, we would like to evaluate cardiometabolic risk factors and the correlation between body mass index, vitamin D stores and inflammatory cytokines.

In an observed, randomized controlled trial over 6 months we will provide observed vitamin D supplementation or placebo to healthy obese and overweight adolescents and measure changes in inflammatory markers, lipids, blood pressure, and mean blood sugars. We hypothesize that administration of vitamin D to these patients will improve their inflammatory profile and cardiometabolic risk factors (blood glucose, blood pressure, and lipid profile).

DETAILED DESCRIPTION:
Supplementation with vitamin D at 150,000 IU every 3 months failed to increase serum 25-hydroxy vitamin D (25OHD) or alter inflammatory markers and lipids in overweight and obese youth. Further studies are needed to establish the dose of vitamin D required to increase 25OHD and determine potential effects on metabolic risk factors in obese teens.

During the course of the study, blood pressure removed from the prespecified outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 11 years to 17.99 years old
2. BMI: 85 percentile for age and gender

Exclusion Criteria:

1. Patients who currently receive:

   * vitamin D supplementation >= 400 IU/day
   * daily glucocorticoids or anti-epileptics
2. Patients who currently have or history of:

   * 25-OH vitamin D level < 10 ng/ml or > 60 ng/ml
   * rickets
   * diabetes mellitus
   * liver or kidney disease
   * malabsorptive disorders
   * genetic syndromes associated with obesity (i.e. Prader-Willi)
   * lactose deficiency or insufficiency
   * galactosemia

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Bachrach, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Shah S, Wilson DM, Bachrach LK. Large Doses of Vitamin D Fail to Increase 25-Hydroxyvitamin D Levels or to Alter Cardiovascular Risk Factors in Obese Adolescents: A Pilot Study. J Adolesc Health. 2015 Jul;57(1):19-23. doi: 10.1016/j.jadohealth.2015.02.006. Epub 2015 Apr 11. PMID 25873553

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: Subjects were assigned to receive two observed doses of vitamin D2 (150,000 IU ergocalciferol, Barr Laboratories and Winthrop (Sanofi-Aventis)), given at baseline and 12 weeks. Capsules were packaged by the hospital's clinical trial pharmacist and were administered by study staff blinded to group assignments.
  Intervention: Height, weight, and BMI were obtained at baseline, 12 weeks and 24 weeks
  Drisdol (Ergocalciferol) Vitamin D2: Ergocalciferol 150,000 IU every 12 weeks for total of 24 weeks.
- Placebo: Subjects were assigned to receive two observed doses of placebo, given at baseline and 12 weeks. Capsules were packaged by the hospital's clinical trial pharmacist and were administered by study staff blinded to group assignments.
  Interventions: Height, weight, and BMI were obtained at baseline, 12 weeks and 24 weeks
  Placebo: Placebo pill - 3 pills every 12 weeks for total of 24 weeks
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 20 | 20
Completed | 14 | 17
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 15.1 [12.4 to 17.6] | 13.6 [11.2 to 16.8] | 14.35 [11.2 to 17.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 8 | 12 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
BMI [Mean (Full Range); unit: kg/m^2] | 36 [25.33 to 48.72] | 31 [23.47 to 41.3] | 33.22 [23.47 to 48.72]
25OH vitamin D [Mean (Full Range); unit: ng/mL] | 19.4 [10 to 30] | 24.2 [12 to 59] | 21.8 [10 to 59]

OUTCOME MEASURES:

1. Primary Outcome: 25OH Vitamin D
Description: Primary outcome is serum 25OH vitamin D concentrations
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
ng/mL
  Baseline | 19.6 (1.4) | 25.8 (2.6)
  Week 24 | 20.1 (0.9) | 24.6 (2.0)

2. Secondary Outcome: Triglycerides at Baseline and Week 24
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
mg/dL
  Baseline | 106 (20) | 99 (13)
  Week 24 | 114 (19) | 99 (11)

3. Secondary Outcome: High-density Lipoprotein (HDL) at Baseline and Week 24
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
mg/dL
  Baseline | 41 (3) | 46 (3)
  Week 24 | 41 (2) | 47 (3)

4. Secondary Outcome: Hemoglobin A1C (HgbA1c) at Baseline and Week 24
Description: HbgA1c is a test to measure of the glucose (blood sugar) level over the past 2-3 months.
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
Percentage of glycosylated hemoglobin
  Baseline | 5.4 (0.1) | 5.3 (0.1)
  Week 24 | 5.4 (0.1) | 5.3 (0.1)

5. Secondary Outcome: Interleukin-6 (IL-6) at Baseline and Week 24
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
pg/mL
  Baseline | 1.0 [0.6 to 1.3] | 0.7 [0.4 to 1.3]
  Week 24 | 1.0 [0.7 to 1.7] | 0.7 [0.4 to 1.2]

6. Secondary Outcome: Interleukin-10 (IL-10) at Baseline and Week 24
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
pg/mL
  Baseline | 1.7 [0.8 to 2.2] | 2.0 [0.8 to 4.6]
  Week 24 | 1.7 [0.7 to 4.1] | 2.3 [1.2 to 4.6]

7. Secondary Outcome: Tumor Necrosis Factor-alpha (TNF-α) at Baseline and Week 24
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
pg/mL
  Baseline | 6.0 [4.9 to 8.7] | 7.2 [6.4 to 7.7]
  Week 24 | 6.9 [5.5 to 8.0] | 7.5 [6.5 to 8.2]

8. Secondary Outcome: C-reactive Protein (CRP) at Baseline and Week 24
Description: Outcome was assessed using high-sensitivity C-reactive protein (hs-CRP) test.
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
mg/L
  Baseline | 4.0 (1.0) | 2.2 (0.5)
  Week 24 | 4.3 (0.9) | 2.3 (0.6)

9. Secondary Outcome: Adiponectin at Baseline and Week 24
Time Frame: Baseline; Week 24
Population: Patients who completed the study were analyzed.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 14 | 17
pg/mL
  Baseline | 4.8 [3.4 to 6.7] | 7.2 [3.6 to 8.8]
  Week 24 | 5.9 [3.6 to 8.9] | 7.3 [4.3 to 11.2]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D (N=20) | Placebo (N=20)
Hypercalcemia (Endocrine disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes